CLINICAL TRIAL: NCT05174481
Title: Forecasting ED Overcrowding With Statistical Methods: A Prospective Validation Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ed-pro
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Emergencies
Keywords: emergency department; overcrowding; forecasting; artificial intelligence; deep learning
MeSH Terms: conditions — Emergencies; Crowding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Early warning system for emergency department overcrowding — In this study, no interventions are performed.

SUMMARY:
The aim of this study is to prospectively validate statistical forecasting tools that have been widely used retrospectively in forecasting ED overcrowding

DETAILED DESCRIPTION:
Emergency department (ED) overcrowding is a chronic international issue that has been repeatedly associated with detrimental treatment outcomes such increased 10-day-mortality. Forecasting future overcrowding would enable pre-emptive staffing decisions that could alleviate or prevent overcrowding along with its detrimental effects.

Over the years, several predictive algorithms have been proposed ranging from generalized linear models to state space models and, more recently, deep learning algorithms. However, the performance of these algorithms has only been reported retrospectively and the clinically significant accuracy of these algorithms remains unclear.

In this study the investigators aim to investigate the accuracy of the previously reported ED forecasting algorithms in a prospective setting analogous to the way these tools would be used if used implemented as a decision-support system in a real-life clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting in the Emergency Department

Exclusion Criteria:

* No exclusion criteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Tampere University Hospital is an academic hospital located in Tampere, Finland. It serves a population of 535,000 in the Pirkanmaa Hospital District and, as a tertiary hospital, an additional population of 365,700 and provides level 1 trauma centre capabilities.
Sampling Method: Non-Probability Sample
Enrollment: 160000 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Next day overcrowding | 24 hours
  A day is defined as overcrowded if daily peak occupancy exceeds 80 patients, and severely overcrowded if daily peak occupancy exceeds 100 patients.

SECONDARY OUTCOMES:
Number of hourly arrivals in the ED 24 hours ahead | 24 hour
Hourly occupancy in the ED 24 hours ahead | 24 hour
Number of daily arrivals in the ED 7 days ahead | 24 hour
Daily peak occupancy in the ED 7 days ahead | 24 hours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gul M, Celik E. An exhaustive review and analysis on applications of statistical forecasting in hospital emergency departments. Health Syst (Basingstoke). 2018 Nov 19;9(4):263-284. doi: 10.1080/20476965.2018.1547348. PMID 33354320
- [Background] Richardson DB. Increase in patient mortality at 10 days associated with emergency department overcrowding. Med J Aust. 2006 Mar 6;184(5):213-6. doi: 10.5694/j.1326-5377.2006.tb00204.x. PMID 16515430